CLINICAL TRIAL: NCT02389270
Title: Age and Daytime Variations in Urinary Neurotrophin Levels in Healthy Children Without Lower Urinary Tract Symptoms
Brief Title: Urinary Neurotrophin Levels in Healthy Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital Zagreb (Other)
Responsible Party: Sponsor
Other Study IDs: pOAB-CHZ-00
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Overactive Bladder
Keywords: Neurotrophins; Nerve Growth Factor; Brain-Derived Neurotrophic Factor; Urinary Biomarkers; Children
MeSH Terms: conditions — Urinary Bladder, Overactive; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine ultrafiltrate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy children: Healthy children without lower urinary tract diseases, history of urinary tract infection, chronic diseases, anomalies of urinary or genital tract, and remarkable clinical examination.

SUMMARY:
The aim of this study is to analyse urinary neurotrophin levels in healthy children. Urine samples will be collected at 3 different times of day (morning, noon, and evening) at urge sensation from all age groups of children who gained bladder control, i.e. from 3-18 years of age. Urinary levels of nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF) normalised to urinary creatinine will be analysed. Age and daytime related variations will be reported for both boys and girls. These results will contribute to understanding the role of neurotrophins in the physiology of lower urinary tract and pathophysiology of idiopathic and secondary hyperactive bladder in children.

ELIGIBILITY:
Inclusion Criteria:

* 3-18 years of age
* a unremarkable clinical examination
* a normal voiding pattern
* a minimum of 3 micturitions per day
* informed oral and written consent from the child and both parents/legal guardian

Exclusion Criteria:

* history of urinary tract infection
* diseases of central or peripheral nerve system
* anomalies of lumbosacral region
* chronic diseases
* operative procedures or anomalies of urinary or genital tract
* lower urinary tract symptoms
* constipation
* hypercalcuria
* urolithiasis, depression, eating disorders or cardio-metabolic diseases
* prior use of anticholinergic treatment

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We will include a group of healthy children recruited from a primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of urinary nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF) normalised to urinary creatinin | Collection of urine samples and analysis will take approximately 6 months.
  We will collect urine samples from healthy children without lower urinary tract symptoms and analyse urine concentrations of neurotrophins (NGF and BDNF) normalised to urinary creatinin in order to report its normal age- and daytime-related variations.

CONTACTS AND LOCATIONS:
Overall Officials: Slaven Abdovic, MD, PhD, Principal Investigator — Children's Hospital Zagreb

IPD SHARING:
Plan to Share IPD: Undecided